CLINICAL TRIAL: NCT06341465
Title: Investigation of the Effects of Exercise and Kinesiological Taping on Spinal Deformities
Brief Title: Investigation of the Effects of Exercise and Kinesiological Taping on Spinal Deformities and Serum Markers in Individuals With Scoliosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Birgül Dıngırdan, Research Assisstant, Sakarya Applied Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HÜ- FTR- BD- 3
Record Dates: First submitted 2024-03-01; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Scoliosis; Scoliosis Idiopathic; Musculoskeletal Deformity
Keywords: Scoliosis; Exercise
MeSH Terms: conditions — Scoliosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 3 groups. Schroth exercise group (n=19), schroth exercise and kinesiological taping group (n=19), healthy people (n=19).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group (Experimental): For 12 weeks, participants will receive rotational breathing, correction techniques, positioning, mobilization, and three-dimensional exercises specific to their curvature twice a week.
  Interventions: Other: Just Exercise
- Exercise and taping group (Experimental): For 12 weeks, participants will schroth exercises including receive rotational breathing, correction techniques, positioning, mobilization and three dimensional exercises specific to their curvature and kinesiological taping. Kinesiological taping will be applied as a tone enhancer or tone reducer according to the concave and convex sides of the curve.
  Interventions: Other: Exercise; Other: Taping
- Healthy people (No Intervention): Healthy individuals without scoliosis will be included.

INTERVENTIONS:
Other: Just Exercise — Schroth exercises are including rotational breathing, correction techniques, positioning, mobilization, and three-dimensional exercises specific to their curvature.
  Arms: Exercise group
Other: Exercise — Schroth exercises are including rotational breathing, correction techniques, positioning, mobilization, and three-dimensional exercises specific to their curvature.
  Arms: Exercise and taping group
Other: Taping — Kinesiological taping will be applied as a tone enhancer or tone reducer according to the the concave and convex sides of the curve.
  Arms: Exercise and taping group

SUMMARY:
The aim of this study is to investigate the effects of Schroth exercises and kinesiological taping on spinal deformities and serum markers in young adults with scoliosis. The study will include young adults aged 18-21 with scoliosis. A total of 57 participants will be included in the study. Out of 57 participants, 38 have scoliosis, and 19 are healthy. 38 participants will be randomly divided into 2 groups. One group (n=19) will receive only Schroth exercises, and the other group (n=19) will receive both Schroth exercises and kinesiological taping. The laboratory analyses of proteins associated with autophagy (Beclin-1, LC3, and ATG3) and bone-cartilage metabolism (COMP and MMP-3) will be conducted in the Biomedical Engineering Laboratory of our university. Trunk rotation will be assessed using the Adams Forward Bend Test with scoliometer, quality of life will be evaluated with the SRS-22 Quality of Life questionnaire and Quality of life profile for spinal deformities questionnaire, perception of deformity will be measured using the Walter Reed Visual Assessment Scale, and Cobb angles will be evaluated from anterior-posterior X-ray images.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of Schroth exercises and kinesiological taping on spinal deformities and serum markers in young adults with scoliosis. The study will include young adults aged 18-21 with scoliosis. A total of 57 participants will be included in the study. Out of 57 participants, 38 have scoliosis, and 19 are healthy. 38 participants will be randomly divided into 2 groups. One group (n=19) will receive only Schroth exercises, and the other group (n=19) will receive both Schroth exercises and kinesiological taping. The laboratory analyses of proteins associated with autophagy (Beclin-1, LC3, and ATG3) and bone-cartilage metabolism (COMP and MMP-3) will be conducted in the Biomedical Engineering Laboratory of our university. Schroth exercises will be administered to both groups twice a week for 12 weeks. Kinesiological taping will be applied twice a week to the group receiving both Schroth exercises and kinesiological taping. Pre-treatment evaluations will include assessments of Cobb angles, trunk rotation, serum markers, quality of life and perception of deformity. Post treatment evaluations will include assessments of trunk rotation, cobb angles, serum markers, quality of life and perception of deformity.

ELIGIBILITY:
Inclusion Criteria:

* The individuals who agree to the study conditions and will continue with the treatment protocol.
* 18-21 years
* Individuals with scoliosis

Exclusion Criteria:

* Individuals with metabolic problems such as diabetes, thyroid issues, kidney problems, etc.
* Individuals with joint diseases such as septic arthritis, viral arthritis, rheumatoid arthritis, etc.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-04-04 (Estimated); Primary Completion 2024-07-04 (Estimated); Study Completion 2024-07-04 (Estimated)

PRIMARY OUTCOMES:
Trunk rotation | At the beginning of the study and three months later
  This method assesses spinal rotation caused by scoliosis. Individuals were asked to stand with their feet together and shoulders width apart, and then to bend forward. Rotation degrees were measured using a scoliometer.
Cobb angles | At the beginning of the study and three months later
  At the beginning and end of the study, participants will have their Cobb angle evaluated from anterior-posterior and posterior-anterior X-ray images.
Serum markers | At the beginning of the study and three months later
  The laboratory analyses of proteins associated with autophagy (Beclin-1, LC3, and ATG3) and bone-cartilage metabolism (COMP and MMP-3) will be conducted in the Biomedical Engineering Laboratory of our university.

SECONDARY OUTCOMES:
Quality of life with scoliosis people | At the beginning of the study and three months later
  The Scoliosis Research Society developed the SRS-22 scale, which is widely accepted for assessing the health-related quality of life in scoliosis patients. Quality of life will be assessed using the SRS-22 questionnaire. The SRS-22 scale consists of 22 questions and 5 subgroups. The subgroups include pain, general appearance (image), spinal function, mental health, and satisfaction with treatment. Scores obtained from each subgroup range from 5 to 25 for pain, general appearance (image), and spinal function, and from 2 to 10 for satisfaction with treatment. Scores are calculated by assigning a response value to each of the 22 questions within a 5-point rating scale. Each statement contains responses ranging from negative to positive. The most negative response receives 1 point, while the most positive receives 5 points. Higher scores on the scale indicate an increase in quality of life, while lower scores indicate a decrease.
Body image assessment | At the beginning of the study and three months later
  Body image assessment will be assessed using the Walter Reed Visual Assessment Scale. WRVAS is a scale developed to evaluate the physical deformity in individuals with scoliosis and the effectiveness of treatment in improving body deformities. It consists of visual representations representing spinal curvature, rib prominence, prominence of the waist, positional relationship of the head-thoracic cage-pelvis, relationship of the head to the pelvis, shoulder level, and scapular rotation. Each deformity in the visuals is scored from a minimum of "1" to a maximum of "5," with higher scores indicating a higher perceived deformity.

IPD SHARING:
Plan to Share IPD: Undecided